CLINICAL TRIAL: NCT07307443
Title: A Phase II Clinical Trial of Anlotinib in Combination With Platinum-based Chemotherapy in Patients With SMARCA4-Deficient, Locally Advanced or Metastatic Lung Cancer.
Brief Title: A Phase II Study of Anlotinib and Platinum-Based Chemotherapy in Patients With SMARCA4-Deficient, Locally Advanced or Metastatic Lung Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhijie Wang (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor-Investigator, Zhijie Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5896
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: SMARCA4-Deficient Tumor; Locally Advanced or Metastatic Lung Cancer
Keywords: SMARCA4-Deficient Locally advanced or Metastatic Lung Cancer; first line therapy; combination therapy; Anlotinib; Platinum-based chemotherapy
MeSH Terms: conditions — Lung Neoplasms | interventions — anlotinib; 130-nm albumin-bound paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combined treatment group (Experimental): This study evaluates a first-line treatment for locally advanced or metastatic SMARCA4-deficient lung cancer, combining Anlotinib-an oral multi-target tyrosine kinase inhibitor that primarily inhibits tumor angiogenesis-with platinum-based chemotherapy. The rationale for this combination is to integrate potent anti-angiogenic therapy with standard cytotoxic chemotherapy, aiming to address the limited efficacy of current standard therapies in this aggressive molecular subset.
  Patients receive the combination of Anlotinib and platinum-doublet chemotherapy for 4-6 induction cycles, followed by Anlotinib monotherapy as maintenance treatment until disease progression or unacceptable toxicity. This design aims to maximize disease control while balancing long-term treatment tolerability.
  No prior prospective clinical studies have specifically evaluated this regimen in patients with SMARCA4-deficient NSCLC confirmed by BRG1 protein loss.
  Interventions: Drug: Anlotinib, nab-paclitaxel, carboplatin

INTERVENTIONS:
Drug: Anlotinib, nab-paclitaxel, carboplatin — Participants will receive Anlotinib (12 mg, orally, once daily on days 1-14) in combination with nab-paclitaxel (260 mg/m², IV, administered as a single dose on day 1 or split between days 1 and 8) and carboplatin (AUC=4-5, IV, day 1) every 21 days for 4-6 induction cycles. Dose adjustments may be made based on clinical judgment and tolerability.
  Patients who do not experience disease progression or intolerable toxicity following the induction phase will proceed to maintenance therapy with Anlotinib monotherapy (12 mg, orally, once daily on days 1-14 every 21 days).
  Treatment will continue until disease progression, unacceptable toxicity, consent withdrawal, investigator decision, loss to follow-up, death, or meeting other protocol-defined criteria for discontinuation.
  The maximum duration of Anlotinib treatment is 24 months. Beyond this period, continuation will be at the investigator's discretion based on an individual benefit-risk assessment.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of combining Anlotinib with platinum-based chemotherapy for treating locally advanced or advanced lung cancer in patients whose tumors are characterized by SMARCA4 deficiency, as evidenced by the loss of BRG1 protein via immunohistochemistry (IHC). It will also learn about the safety of this combination treatment.

The main questions it aims to answer are:

1. How long can this treatment delay the worsening of the cancer (Progression-Free Survival, PFS)?
2. What side effects or medical problems do participants have when taking this combination? This is a single-arm study, meaning all participants will receive the same investigational combination therapy. Researchers will monitor how well the cancer responds and compare the results to historical data from similar patients who received other treatments.

Participants will:

1. Receive treatment in 21-day cycles: take Anlotinib pills on days 1-14 of each cycle and receive platinum-based chemotherapy by intravenous infusion on day 1 (or days 1 and 8).
2. Undergo regular clinic visits for imaging scans (like CT scans), blood tests, and physical examinations to check the cancer's status and their overall health.
3. Complete questionnaires about their quality of life.
4. Provide tumor tissue and blood samples for exploratory research to understand which patients might benefit most from this treatment.

Treatment will continue until the cancer worsens, side effects become intolerable, the participant decides to withdraw, or the study ends.

DETAILED DESCRIPTION:
SMARCA4-deficient non-small cell lung cancer (NSCLC) is a distinct and highly aggressive molecular subtype, characterized by inactivating mutations or loss of the SMARCA4 gene, which encodes the BRG1 protein. It constitutes approximately 5-10% of all NSCLC cases. Patients typically present with advanced-stage disease at diagnosis and exhibit a notoriously poor prognosis, with historical median overall survival (mOS) often ranging from 4 to 7 months. Current standard first-line therapies, including immune checkpoint inhibitor (ICI) combinations, have shown limited and inconsistent efficacy in this specific population, creating a significant unmet medical need.

Therapeutic options for SMARCA4-deficient NSCLC remain an area of active investigation. While platinum-doublet chemotherapy forms the backbone of treatment, the added benefit of ICIs is ambiguous. Large retrospective analyses suggest that tumors harboring SMARCA4 alterations may derive less benefit from frontline chemoimmunotherapy compared to wild-type tumors, highlighting the intrinsic resistance mechanisms and unique tumor microenvironment of this subtype. Therefore, exploring novel combination strategies beyond conventional immunotherapy is critical.

Anlotinib is an orally administered, multi-targeted tyrosine kinase inhibitor that potently inhibits key angiogenesis pathways (VEGFR, PDGFR, FGFR) as well as tumor proliferation pathways (c-Kit, RET). It is approved in China for later-line treatment of advanced NSCLC. Beyond its anti-angiogenic effects, preclinical and clinical evidence suggests that Anlotinib may modulate the tumor immune microenvironment and synergize with chemotherapy to enhance anti-tumor activity. The rationale for combining Anlotinib with platinum-based chemotherapy in SMARCA4-deficient NSCLC is multi-faceted: 1) to provide a robust cytotoxic backbone; 2) to simultaneously inhibit tumor angiogenesis, a potential driver of aggressiveness; and 3) to potentially re-sensitize or circumvent the relative immunotherapy resistance observed in this subtype.

To date, no prospective clinical trial data exist on the use of Anlotinib combined with platinum-based chemotherapy as a first-line treatment for SMARCA4-deficient NSCLC. This phase II, single-arm, open-label study is designed to prospectively evaluate the efficacy and safety of this novel combination regimen in patients with locally advanced or metastatic SMARCA4-deficient NSCLC, confirmed by immunohistochemical loss of BRG1 protein.

The primary objective is to assess progression-free survival (PFS). Secondary objectives include objective response rate (ORR), disease control rate (DCR), duration of response (DoR), overall survival (OS), safety profile, and health-related quality of life (HRQoL). Exploratory biomarker analyses on tumor tissue and blood samples will investigate molecular features of the tumor and its microenvironment to identify potential predictors of response and resistance.

This study aims to generate the first prospective evidence for a targeted-chemotherapy combination in this challenging disease, potentially offering a new and effective first-line treatment strategy for patients with SMARCA4-deficient NSCLC.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL the following criteria to be eligible for trial participation:

1. Voluntary participation and provision of written informed consent.
2. Age ≥ 18 years.
3. Life expectancy ≥ 3 months.
4. Diagnosed with unresectable, locally advanced (Stage IIIB) or metastatic (Stage IV) lung cancer not amenable to curative radiotherapy.
5. Tumor confirmed by immunohistochemistry (IHC) to be deficient in the BRG1 protein (encoded by the SMARCA4 gene).
6. No prior systemic anti-cancer therapy.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
8. Willing and able to provide archival or fresh tumor tissue samples from primary or metastatic sites for biomarker analysis. Enrollment may be considered after investigator assessment if tissue is unavailable, provided all other criteria are met.
9. At least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
10. Adequate organ and bone marrow function as defined by the following laboratory values (within screening period):

10.1. Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L. 10.2. Platelet count ≥ 100 × 10⁹/L. 10.3. Hemoglobin ≥ 90 g/L (without blood transfusion within 14 days). 10.4. Serum creatinine ≤ 1 × Upper Limit of Normal (ULN) OR estimated creatinine clearance > 50 mL/min (Cockcroft-Gault formula).

10.5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN if liver metastases are present).

10.6. Total bilirubin ≤ 1.5 × ULN (For subjects with Gilbert's syndrome, total bilirubin must be < 51.3 µmol/L).

10.7. Prothrombin time (PT), activated partial thromboplastin time (APTT), and International Normalized Ratio (INR) ≤ 1.5 × ULN (for subjects not receiving anticoagulant therapy).

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded from the trial:

1. Pathological diagnosis containing a small cell carcinoma component.
2. Symptomatic brain metastases.
3. Leptomeningeal carcinomatosis.
4. Failure to recover from acute toxicities of prior anti-cancer therapy to ≤ Grade 1 per NCI CTCAE v5.0 or to baseline levels specified in the inclusion criteria (excluding alopecia or fatigue) within 4 weeks prior to the first dose.
5. Conditions that compromise intravenous access or oral drug administration (e.g., inability to swallow, chronic diarrhea, intestinal obstruction); OR unwillingness or inability to undergo a repeat biopsy or provide sufficient tissue samples for comprehensive analysis (whole-exome sequencing, transcriptome sequencing, multiplex fluorescence immunohistochemistry).
6. Failure to recover from adverse reactions of prior therapies to ≤ Grade 1 per CTCAE v5.0, except for toxicities deemed by the investigator to pose no safety risk (e.g., Grade 2 alopecia, Grade 2 peripheral neuropathy, Grade 2 anemia, non-clinically significant and asymptomatic laboratory abnormalities, or stable hypothyroidism on hormone replacement therapy).
7. Major surgical procedure, significant traumatic injury within 4 weeks prior to the first dose, or anticipated need for major surgery during the study treatment period (unless specified in the protocol); OR presence of non-healing wounds or fractures. (Major surgery is defined as Grade 3 or higher according to the National Surgery Classification Catalog 2022 edition).
8. Any arterial or venous thromboembolic event (e.g., cerebrovascular accident, transient ischemic attack, deep vein thrombosis, pulmonary embolism) within 6 months prior to the first dose; OR any bleeding or hemorrhagic event ≥ Grade 3 per CTCAE v5.0 within 4 weeks prior to the first dose.
9. Poorly controlled active viral hepatitis. Eligible subjects meeting the following criteria may be screened:

   9.1 HBsAg-positive subjects must have HBV DNA < 2000 IU/mL (or 1×10⁴ copies/mL) OR have received at least 1 week of anti-HBV therapy prior to study initiation with at least a 10-fold (1-log) reduction in viral load, AND agree to receive continuous anti-HBV therapy throughout the study.

   9.2 HCV-infected subjects (HCV Ab or HCV RNA positive) must be in a stable condition as judged by the investigator OR be receiving approved antiviral therapy at enrollment and willing to continue it during the study.
10. History of psychotropic substance abuse with inability to abstain, or presence of psychiatric disorders.
11. Prior or planned allogeneic bone marrow transplantation or solid organ transplantation.
12. History of hepatic encephalopathy.
13. Significant cardiovascular disease, including any of the following:

    13.1 Cardiac insufficiency ≥ Class II per New York Heart Association (NYHA) criteria OR left ventricular ejection fraction (LVEF) < 50% on echocardiography.

    13.2 History of clinically significant ventricular arrhythmia (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes) OR arrhythmia requiring ongoing antiarrhythmic medication.

    13.3 Unstable angina. 13.4 Myocardial infarction within the past 12 months. 13.5 QTcF interval > 450 msec for males or > 470 msec for females (if abnormal, the average of three consecutive readings taken at least 2 minutes apart).

    13.6 Personal or family history of congenital long QT syndrome. 13.7 History of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolism within 3 months prior to randomization (thrombosis related to implanted ports/catheters or superficial thrombophlebitis are not considered "severe").

    13.8 Current use or recent use (within 7 days prior to treatment initiation) of aspirin (>325 mg/day), dipyridamole, ticlopidine, clopidogrel, or cilostazol.
14. Poorly controlled concurrent illnesses, such as:

    14.1 Serious infection within 4 weeks prior to treatment initiation requiring hospitalization; OR therapeutic oral/intravenous antibiotics within 2 weeks prior to treatment initiation (prophylactic antibiotic use is permitted, e.g., for urinary tract infection or COPD).

    14.2 Symptomatic congestive heart failure (NYHA Class II-IV) OR symptomatic/poorly controlled arrhythmia.

    14.3 Other active malignancy diagnosed within the past 5 years, except for curatively treated non-melanoma skin cancer, basal/squamous cell carcinoma, or carcinoma in situ (e.g., breast, cervix, bladder) with no evidence of recurrence.

    14.4 Suspected or confirmed acute promyelocytic leukemia (for patients with acute myeloid leukemia).

    14.5 Current carcinomatous meningitis or spinal cord compression. 14.6 Poorly controlled hypertension. 14.7 Symptomatic intrinsic lung disease. 14.8 Any arterial thromboembolic event within 6 months prior to enrollment, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack.

    14.9 Significant malnutrition requiring intravenous nutritional support, unless corrected and stable for ≥ 4 weeks prior to the first dose.

    14.10 Tumor invasion of adjacent vital organs or major blood vessels (e.g., mediastinal great vessels, superior vena cava, trachea, esophagus), or risk of esophageal-tracheal or esophageal-pleural fistula.

    14.11 History of esophageal or tracheal stent implantation. 14.12 Any other acute/chronic illness or laboratory abnormality that, in the investigator's judgment, increases risk associated with study participation or drug administration, OR interferes with the interpretation of study results.

    14.13 History of gastrointestinal perforation and/or fistula within 6 months prior to enrollment.

    14.14 Uncontrolled third-space effusions requiring repeated drainage (e.g., pleural, peritoneal, pericardial effusion). Subjects not requiring drainage or stable for 3 days after stopping drainage may be eligible.
15. Active gastrointestinal diseases or other conditions that may significantly affect drug absorption, metabolism, or excretion, including but not limited to: malabsorption syndrome, inflammatory bowel disease, partial or complete intestinal obstruction, gastrectomy, or small bowel resection.
16. Severe underlying pulmonary disease or history thereof, such as moderate to severe chronic obstructive pulmonary disease (COPD), history of interstitial lung disease (ILD), drug-induced ILD, acute or chronic infectious pneumonia, or lung transplantation.
17. Pregnant or lactating women.
18. Concurrent participation in another interventional clinical trial, or an observational (non-interventional) clinical study, or being in the follow-up phase of an interventional study.
19. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
20. Major surgical procedure (as defined by the investigator, e.g., craniotomy, thoracotomy, laparotomy, vascular intervention) within 4 weeks prior to the first study drug dose, OR presence of unhealed wounds, ulcers, or fractures. Note: Palliative local surgery for isolated lesions is acceptable.
21. HIV infection (HIV 1/2 antibody positive).
22. Known active syphilis infection or active tuberculosis.
23. Documented history of psychiatric disorder requiring medication.
24. History of drug abuse or substance addiction.
25. Any other condition that, in the judgment of the investigator, may affect study results, interfere with the subject's participation in the entire study process, or render the subject unsuitable for participation, including but not limited to existing or past medical conditions, treatments, laboratory abnormalities, or unwillingness to comply with study procedures and requirements.
26. Use of any other investigational drug or therapy within 4 weeks prior to the first study dose.
27. Use of any Chinese herbal medicine with anti-tumor activity within 2 weeks prior to initiation of study treatment.
28. History of other malignancies (excluding non-melanoma skin cancer and carcinoma in situ of the bladder, stomach, colon, endometrium, cervix/dysplasia, melanoma, or breast), unless the subject has been in complete remission for at least 2 years prior to enrollment and requires no other treatment during the study.
29. Planned administration or administration of a live vaccine within 28 days prior to the first study dose.
30. Known hypersensitivity or intolerance to the study drug(s) or any of their excipients.
31. Any other condition that, in the investigator's opinion, makes the subject unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to the end of monitoring at 2 years.
  PFS is defined as the time from the first dose of study treatment to the first documentation of disease progression according to RECIST v1.1 (as assessed by investigators) or death from any cause, whichever occurs first. Subjects who are alive without progression at the time of analysis will be censored at the date of the last tumor assessment.

SECONDARY OUTCOMES:
Overall Survival (OS) | From enrollment to the end of monitoring at 2 years.
  OS is defined as the time from the first dose of study treatment to death from any cause. Subjects who are alive at the time of analysis will be censored at the date of last follow-up.
Objective Response Rate (ORR) | From enrollment to the end of monitoring at 2 years.
  ORR is defined as the proportion of subjects who achieve a complete response (CR) or partial response (PR) as per RECIST v1.1.
Duration of Response (DoR) | From enrollment to the end of monitoring at 2 years.
  DoR is defined as the time from the first documentation of CR or PR to the first documentation of disease progression or death.
Disease Control Rate (DCR) | From enrollment to the end of monitoring at 2 years.
  DCR is defined as the proportion of subjects who achieve CR, PR, or stable disease (SD) as their best overall response.
The incidence of adverse events | From enrollment to the end of monitoring at 2 years
  Incidence, nature, and severity of adverse events (AEs), graded according to NCI-CTCAE v5.0, including immune-related AEs and serious AEs.
Health-Related Quality of Life (HRQoL) | From enrollment to the end of monitoring at 2 years
  HRQoL will be assessed using the 36-Item Short Form Survey (SF-36v2), focusing on both physical (PCS) and mental (MCS) component summary scores.

OTHER OUTCOMES:
Biomarker Discovery | From enrollment to the end of monitoring at 2 years
  Collection of tumor tissue and peripheral blood samples at baseline and disease progression for multi-omics analysis (e.g., DNA, RNA) to characterize tumor and microenvironment features and identify potential biomarkers of treatment efficacy and toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No